CLINICAL TRIAL: NCT02814968
Title: A Phase 2, Open-label, Single-arm, Efficacy and Imaging Study of Oral Enzalutamide in Chemo-Naïve Patients With Progressive Prostate Cancer Who Have Failed Androgen Deprivation Therapy (Castration-resistant Prostate Cancer Patients)
Brief Title: PET/CT and WB MRI for Staging and Response in CRPC Patients Receiving Enzalutamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The European Uro-Oncology Group (Other)
Collaborators: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT Number 2014-001161-27
Record Dates: First submitted 2016-06-18; First posted 2016-06-28 (Estimated); Last update posted 2022-04-14 (Actual); Status verified 2021-02

CONDITIONS: Prostate Cancer Metastatic
Keywords: Castration-resistant prostate cancer; Enzalutamide; Imaging; PET/CT; Whole body MRI; Circulating tumour cells; Cell-free tumour DNA
MeSH Terms: interventions — enzalutamide

ARMS (1):
- Single arm (Experimental): Subjects will receive 1 dd 160 mg Enzalutamide orally continuously until progressive disease occurs. Serial PSA measurements, PET/CT scans, Whole Body MRI, bone scans will be performed to assess metastatic tumour load, progressive disease and response to treatment.
  Interventions: Drug: Enzalutamide; Device: 18-FDG PET/CT; Device: Whole body MRI; Device: Bone scan

INTERVENTIONS:
Drug: Enzalutamide
  Other Names: Xtandi
Device: 18-FDG PET/CT
Device: Whole body MRI
Device: Bone scan

SUMMARY:
The aim of the study is to assess the clinical utility of 18F-fluoro-deoxyglucose Positron Emission Tomography (PET)/Computed Tomography (CT) and Whole Body Magnetic Resonance Imaging (MRI) versus conventional bone scan and prostate-specific antigen (PSA) measurements in response prediction to treatment with Enzalutamide in castration-resistant prostate cancer patients.

The study will assess how these 2 imaging modalities perform compared to traditional serial PSA measurements and bone scan in assessing metastatic tumour load, progressive disease and response to treatment with Enzalutamide in castration-resistant prostate cancer patients.

In addition measurements of serially collected circulating tumour cell (CTC) samples, cell-free tumour DNA and RNA will be performed in order to evaluate their predictive value in terms of response measurement.

DETAILED DESCRIPTION:
Castration-resistant prostate cancer patients eligible for 2nd line hormonal treatment will undergo treatment with Enzalutamide (XTANDI). Subjects will receive 1dd 160 mg Enzalutamide orally continuously until progressive disease occurs.

All subjects will undergo 18F-FDG PET/CT scans at baseline, 2 weeks, 2 and 6, 9 and 12 months after starting androgen receptor-directed treatment. All subjects will undergo Whole Body MRI at baseline, 6, 9 and 12 months. Bone scans will be performed at baseline, 3 months, 6 and 12 months. PSA will be measured at baseline and every 4 weeks thereafter until at 12 months. CTC counts and characteristics will be measured at baseline and during Enzalutamide treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 18 years or older;
* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features;
* Ongoing androgen deprivation therapy with a GnRH analogue or bilateral orchiectomy;
* Three consecutive rises of PSA, 1 week apart, resulting in two 50% increases over the nadir, with PSA of at least > 5 ng/mL but preferably >10 ng/mL;
* Progressive disease as defined by rising PSA levels plus by evidence of progressive and measurable soft tissue or bone disease by 18F-FDG PET/CT, Whole Body MRI or both;
* Castrate serum levels of testosterone < 50 ng/dL or < 1.7 nmol/L;
* Anti-androgen withdrawal for at least 6 weeks for bicalutamide, nilutamide or flutamide for at least 6 weeks;
* No prior treatment with cytotoxic chemotherapy;
* Eastern Cooperative Oncology Group (ECOG) score 0-2;
* A life expectancy of at least 12 months;
* Written informed consent.

Exclusion Criteria:

* Severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the patient inappropriate for enrolment;
* Known or suspected brain metastasis or active leptomeningeal disease;
* History of another malignancy within the previous 5 years other than curatively treated non melanomatous skin cancer;
* Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) 2.5 times the upper limit of normal at the Screening visit;
* Creatinine > 177 µmol/L (2 mg/dL) at the Screening visit;
* Hemoglobin <6 mmol/L, White blood cells < 4.0 x10^9/L, platelets < 100 x 10^9/L;
* History of seizure or any condition that may predispose to seizure. Also, history of loss of consciousness or transient ischemic attack within 12 months of enrolment (Day 1 visit);
* Contra-indication for MRI (e.g. pacemaker).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-02; Primary Completion 2020-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) at 6 months | 6 months
  Defined as the time from the date of randomization to the date of radiological progression or death (patients will be followed beyond the fixed time point of 12 months for continued response cq recurrence, but 12 month is the last fixed primary endpoint assessment). Radiological progression is defined by any of the following criteria:
  * Soft tissue lesions: Progressive disease on 18F-FDG PET/CT or MRI by RECIST 1.1. Bone or bone marrow lesions: Progressive disease on PET/CT or MRI as evidenced by new lesions or an increase in size of 25% of the sum of target lesions.
  * Conversion of the 18F-FDG PET signal of the metastases at 2 weeks, 2 or 6 months compared to baseline PET which by comparing it to PFS at 6 and 12 months may be an indicator or drug response. Radiological PFS at 6 months will be compared to a) PET signal conversion and to b) PSA measurements, and changes in number of lesions on the bone scan (conventional work up).
Progression-Free Survival (PFS) at 12 months | 12 months
  Defined as the time from the date of randomization to the date of radiological progression or death (patients will be followed beyond the fixed time point of 12 months for continued response cq recurrence, but 12 month is the last fixed primary endpoint assessment). Radiological progression is defined by any of the following criteria:
  * Soft tissue lesions: Progressive disease on 18F-FDG PET/CT or MRI by RECIST 1.1. Bone or bone marrow lesions: Progressive disease on PET/CT or MRI as evidenced by new lesions or an increase in size of 25% of the sum of target lesions.
  * Conversion of the 18F-FDG PET signal of the metastases at 2 weeks, 2 or 6 months compared to baseline PET which by comparing it to PFS at 6 and 12 months may be an indicator or drug response. Radiological PFS at 12 months will be compared to a) PET signal conversion and to b) PSA measurements, and changes in number of lesions on the bone scan (conventional work up).

SECONDARY OUTCOMES:
Biochemical (PSA) response defined as prostate-specific antigen (PSA) nadir. | 12 months
  Response as PSA nadir.
PSA progression. PSA kinetics measured by PSA doubling time (regular PSA measurements). | 12 months
  PSA doubling time
Progression of bone lesions detected with bone scan according to Prostate Cancer Working Group 2 (PCWG2) criteria. | 6 and 12 months
  Progression of bone lesions
Radiologically confirmed spinal cord compression or pathological fracture due to malignant progression. | 6 and 12 months
  Radiological assessment of spinal cord compression or pathological fracture
Occurrence of Symptomatic Skeletal Events (SSE) evaluated by combination of clinical and radiological assessments | 12 months
  Assessment of external beam radiation therapy to relieve skeletal pain, occurrence of a new symptomatic pathologic bone fracture, spinal cord compression, tumour-related orthopedic surgical intervention or change of anti-neoplastic therapy to treat bone pain
Number of participants with change in CTC measurements correlated to radiological PFS. | 6 and 12 months
  Assessment of radiological PFS
Percent change from baseline in serum concentration of circulating testosterone (T). | 12 months
  Change in circulating testosterone
Percent change from baseline in serum concentration of dihydrotestosterone (DHT). | 12 months
  Change in serum concentration of dihydrotestosterone
Percent change from baseline in serum concentration of sex hormone binding globulin (SHBG). | 12 months
  Changes of SHBG
Percent change from baseline in serum concentration of androstenedione (A). | 12 months
  Changes of androstenedione from baseline
Number of participants with changes in biomarkers of bone turnover correlated to PSA. | 12 months
  Changes in biomarkers
Number of participants with adverse events (AEs) and serious adverse events (SAEs) leading to treatment discontinuation. | 6 and 12 months
  Assessment of AE and SAEs
Time to symptomatic progression (including death due to prostate cancer). | 12 months
  Time to progression
Time to initiation of salvage systemic therapy, including chemotherapy, or palliative radiation. | 12 months
  Time to chemotherapy or palliative radiation.
Quality of life measured by the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire. | 6 and 12 months
  Quality of life assessment
Quality of life measured by the EuroQol 5-Dimension QoL Instrument (EQ-5D). | 6 and 12 months
  Quality of life assessment
Changes in Karnofsky score | 6 and 12 months
  Changes in Karnofsky score
Changes in visual analogue scale (VAS) for tumour-related pain. | 6 and 12 months
  Pain changes from baseline (QoL)
Changes in bone mineral density (BMD) as measured by Dual-energy X-ray absorptiometry (DXA) scan. | 6 and 12 months
  Bone mineral density changes

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Osanto, MD PhD, Study Chair — The European Uro-Oncology Group (EUOG)
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- See also: The European Uro-Oncology Group — http://euog.org/